CLINICAL TRIAL: NCT04620694
Title: Impact of Arterial Cannulation Site on Vasopressor Requirement During Cardiac Surgery: a Monocentric Prospective Cohort Study
Brief Title: Impact of Arterial Cannulation Site on Vasopressor Requirement in Cardiac Surgery
Acronym: ATRAP-GCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0947
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Disease
Keywords: Cardiac surgery; Aortic to radial arterial pressure gradient; Vasopressor
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radial artery cannulation: Patients whom radial artery was cannulated at the beginning of the surgery.
- Aortic cannulation (brachial or femoral artery): Patients whom femoral or brachial artery was cannulated at the beginning of the surgery.
  Active comparator
  Interventions: Device: Choice of arterial cannulation site at the beginning of the surgery

INTERVENTIONS:
Device: Choice of arterial cannulation site at the beginning of the surgery — Choice of arterial cannulation site at the beginning of the surgery is at the discretion of the anesthesia physician.
  Groups: Aortic cannulation (brachial or femoral artery)

SUMMARY:
Choice of arterial cannulation site during cardiac surgery is controversial. Some physicians in our institution prefer radial artery site, others prefer aortic site (via femoral artery or brachial artery). The investigators aim to compare these two strategies for vasopressor requirement. The study hypothesis is that radial artery cannulation is associated with a larger dose of vasopressor due aortic to radial arterial pressure gradient phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Scheduled for cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* More than one arterial cannula at the beginning of the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for cadiac surgery wih cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Intraoperative vasopressor requirement | end of surgery
  Mean intraoperative dosage of Norepinephrine (µg.kg-1.min-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided